CLINICAL TRIAL: NCT03916458
Title: REGISTRY OF COMPLETE RESPONSES TO SUNITINIB IN SPANISH PATIENTS WITH METASTATIC RENAL CELL CARCINOMA (ATILA STUDY)
Brief Title: REGISTRY OF COMPLETE RESPONSES TO SUNITINIB IN SPANISH PATIENTS WITH METASTATIC RENAL CELL CARCINOMA
Acronym: ATILA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181227; ATILA (Other: Alias Study Number)
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-10

CONDITIONS: Carcinoma, Renal Cell
Keywords: Carcinoma, Renal Cell; Disease-Free Survival; Sunitinib; Protein Kinase Inhibitors; Angiogenesis Inhibitors; Prognosis
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with reported metastatic renal cell carcinoma: The subjects have been treatment with sunitinib and they reached complete remission

SUMMARY:
Observational, retrospective, multicentre study in spanish patients with metastatic Renal Cell Carcinoma (mRCC) treated with sunitinib as a first-line treatment (treatment with previous cytokine therapy is accepted) according to clinical practice who obtained a complete response (CR) to treatment in one of these 2 situations:

1. Complete response (CR) obtained exclusively with first-line sunitinib treatment (sunitinib CR).
2. Response obtained after a period of time on treatment with sunitinib in which local treatment was also performed (surgery of the residual metastasis/metastases, radiofrequency ablation or radiotherapy) to achieve the total macroscopic disappearance of the disease, according to the opinion of the physician responsible for the patient (CR + local treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 year-old or over who have been treated for metastatic renal cell carcinoma with sunitinib as first-line treatment (treatment with prior cytokine therapy is accepted) between 2007 and 30 September 2018 and who have obtained as a best treatment response the total remission of the disease in the opinion of the doctor in charge from a clinical, radiological and/or macroscopic point of view. This response must have been reached through two possible strategies:

   A) Systemic treatment with sunitinib alone. B) Treatment with sunitinib and subsequent local treatment for one or more residual lesions that have not responded to the drug (traditional surgery, radiotherapy, SBRT (Stereotactic Body Radiation Therapy)).
2. The duration of CR must have been confirmed with at least 2 consecutive imaging tests, without having a limit in the duration of this response. Although the patient had progressed subsequently, he/she may be included in this registry.
3. Patients from any risk group
4. Tumours of any histology

Exclusion Criteria:

1. Patients treated with another drug other than Sunitinib.
2. Patients with no radiology reports proving CR.
3. Patients with no record of the dose and regimen received with Sunitinib.
4. Patients who achieved complete remission after 30 September 2018.

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population eligible for this study includes any patient with advanced or metastatic renal cell cancer who has been treated with Sunitinib and has achieved CR of the tumour and its metastases at any time during treatment and according to the usual assessment criteria in daily clinical practice, whether it was obtained with sunitinib alone or if a local treatment was needed to eradicate all the lesions: (surgery of the residual metastases, radiofrequency ablation or radiotherapy)
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (31):
- Spain (31):
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital San Juan de Dios, Manresa, Barcelona
  - Hospital Parc Taulí de Sabadell, Sabadell, Barcelona
  - Hospital Universitario Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Infanta Cristina, Parla, Madrid
  - Hospita Virgen de la Salud, Toledo, Madrid
  - Hospital Universitario Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Complexo Hospitalario Universitario de Ferrol, A Coruña
  - Hospital Universitario Infanta Cristina, Badajoz
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant, Barcelona
  - Hospital Clínico de Barcelona, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario de León, León
  - Hospital Universitario Lucus Augusti / Servicio de Oncología Médica, Lugo
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos de Madrid, Madrid
  - Hospital Universitario 12 de octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complexo Hospitalario Universitario de Ourense, Ourense
  - Complejo Asistencial de Segovia, Segovia
  - Hospital de Valme, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] de Velasco G, Alonso-Gordoa T, Rodriguez-Vida A, Anguera G, Campayo M, Pinto A, Ortega EM, Gallardo E, Nunez NF, Garcia-Carbonero I, Reig O, Mendez-Vidal MJ, Fernandez-Calvo O, Cassinello NV, Torregrosa D, Lopez-Martin A, Rosero A, Valiente PG, de Espana CG, Climent MA, Santasusana MD, Sanchez AR, Gonzalez IC, Afonso R, Garcia Del Muro X, Casinello J, Fernandez-Parra EM, Garcia Sanchez L, Afonso J, Polo SH, Asensio U. Long-term Clinical Outcomes of a Spanish Cohort of Metastatic Renal Cell Carcinoma Patients with a Complete Response to Sunitinib. Clin Genitourin Cancer. 2023 Jun;21(3):e166-e174. doi: 10.1016/j.clgc.2022.11.021. Epub 2022 Dec 5. PMID 36610891
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A6181227

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged above or equal to 18 years, with metastatic renal cell carcinoma (mRCC), and who according to the usual evaluation criteria in daily clinical practice obtained a complete response with sunitinib as first-line treatment between 2007 and 30 October 2018, either alone or with subsequent local treatment, were observed retrospectively in this study for a period of 10 months approximately.
Groups:
- Sunitinib: Participants who received sunitinib as first line therapy (treatment with prior cytokine therapy was accepted) in real world clinical practices, between 2007 and 30 October 2018, either alone or with subsequent local treatment (surgery of the residual metastasis/metastases, radiofrequency ablation or radiotherapy) and achieved a complete response were observed in the study. The participants were administered with sunitinib 50 milligrams (mg) capsule orally once daily on a schedule of 4 weeks on treatment followed by 2 weeks off treatment (4/2 regimen) or 2 weeks on treatment followed by 1 week off treatment (2/1 regimen), or with 37.5 mg capsule orally once daily of 4/2 regimen.
Period: Overall Study
Arm/Group | Sunitinib
Started | 62
Completed | 62 (Out of these 62 participants, 2 participants died. But data available before censoring date for these 2 participants were observed and included in results.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who met the inclusion criteria and who did not meet any of the exclusion criteria and received treatment with sunitinib prior to participation in the registry were considered evaluable.
Groups:
- Sunitinib: Participants who received sunitinib as first line therapy (treatment with prior cytokine therapy was accepted) in real world clinical practices, between 2007 and 30 October 2018, either alone or with subsequent local treatment (surgery of the residual metastasis/metastases, radiofrequency ablation or radiotherapy) and achieved a complete response were observed in the study. The participants were administered with sunitinib 50 mg capsule orally once daily on a schedule of 4 weeks on treatment followed by 2 weeks off treatment (4/2 regimen) or 2 weeks on treatment followed by 1 week off treatment (2/1 regimen), or with 37.5 mg capsule orally once daily of 4/2 regimen.
Arm/Group | Sunitinib
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.3 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data was never collected.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Participants With Comorbidities [Count of Participants; unit: Participants] — Comorbidities at baseline included cardiovascular disease, liver disorders, renal failure, autoimmune disease, chronic dermatological disease, obesity, bowel disease and other disease. One participant might have more than 1 comorbidity.
  Participants
    Cardiovascular Disease | 29
    Liver Disorders | 2
    Renal Failure | 5
    Autoimmune Disease | 0
    Chronic Dermatological Disease | 1
    Obesity | 11
    Bowel Disease | 1
    Other Disease | 28
Participants With Number of Metastatic Sites [Count of Participants; unit: Participants] — Here, number of participants were classified according to number of metastatic sites.
  Participants
    1 | 25
    2 | 13
    3 | 7
    4 | 2
    5 | 4
    Greater than (>) 5 | 3
    Data not available | 8
Number of Participants According to Type of Metastatic Sites [Count of Participants; unit: Participants] — Here, number of participants were classified according to type of metastatic sites. One participant might have more than metastatic sites.
  Participants
    Lung | 42
    Liver | 6
    Brain | 2
    Pancreas | 5
    Contralateral Kidney | 2
    Nodes | 23
    Bone | 6
    Muscles, Soft tissues, Vessels and Peritoneum | 8
    Endocrine Glands | 6
Number of Participants Classified According to Tumor Fuhrman Grade [Count of Participants; unit: Participants] — The four-tiered Fuhrman grading evaluates nuclear size, nuclear shape and presence of nucleolar prominence. Grade I - small (=10 micrometer [mcm]) nuclear diameter, round/uniform nuclear shape and absent/inconspicuous nucleoli; Grade II - large (=15 mcm) nuclear diameter, irregular outline nuclear shape and visible at *400 magnification nucleoli; Grade III - Larger (=20 mcm) nuclear diameter, obvious irregular outline nuclear shape and visible and prominent at *100 magnification nucleoli; Grade IV - grade 3 plus bizarre multilobed nuclei +/- spindle cells.
  Participants
    I | 3
    II | 23
    III | 18
    IV | 9
    II and IV | 1
    Data not available | 8
Histological Type of Tumor [Count of Participants; unit: Participants] — Here, number of participants were classified according to type of histology as clear cell, non-clear cell and sarcomatoid.
  Participants
    Clear Cell | 49
    Non-clear Cell | 5
    Sarcomatoid | 7
    Data not available | 1
Pre-treatment Necrosis Percentage [Mean (Standard Deviation); unit: Percentage of Necrosis] — Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Percentage of Necrosis
    number analyzed (Participants) | 13
    (all) | 18.2 (30.4)
Number of Participants With Previous Nephrectomy Status [Count of Participants; unit: Participants] — Here, number of participants were classified according to presence of previous nephrectomy as Yes or No.
  Participants
    Yes | 56
    No | 6
Time Interval From Nephrectomy to Initiation of Sunitinib Treatment [Median (Full Range); unit: Months] — Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Months
    number analyzed (Participants) | 56
    (all) | 15.3 [0.5 to 174.8]
Number of Participants Classified According to Motzer Prognostic Criteria [Count of Participants; unit: Participants] — Motzer prognostic model identified karnofsky performance status(KPS) less than (<)80 at treatment initiation, period from diagnosis to start of treatment for metastatic disease <1 year, anemia, hypercalcemia, elevated lactate dehydrogenase as prognostic factors. Participants were classified into prognosis group: favorable(0 factor), intermediate(1-2 factors), poor(3 or more factors). KPS measured ability of participants with cancer to perform ordinary tasks. KPS scores range: 0 (dead) to 100 (normal, no complaint). High score= participant better able to carry out daily activities. Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 55
    Favorable | 11
    Intermediate | 42
    Poor | 2
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS: measure quality of life of cancer participants on a 0 to 5 scale; 0= fully active, able to carry on all pre-disease performance without restriction; 1= restricted in physically strenuous activity, ambulatory, able to carry out light/ sedentary work; 2= ambulatory, capable of all self-care, unable to carry out any work activity, up >50 % of waking hours; 3= capable of only limited self-care, confined to bed/ chair >50% of waking hours; 4= completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5= dead.
  Participants
    0 | 38
    1 | 22
    2 | 1
    Data not available | 1
Blood Hemoglobin Level [Mean (Standard Deviation); unit: Gram per deciliter] — Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Gram per deciliter
    number analyzed (Participants) | 60
    (all) | 14.0 (3.1)
Corrected Blood Calcium Level [Mean (Standard Deviation); unit: Milligram per deciliter] — Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Milligram per deciliter
    number analyzed (Participants) | 49
    (all) | 9.4 (0.9)
Blood Lactate Dehydrogenase (LDH) Level [Mean (Standard Deviation); unit: Units per liter] — Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Units per liter
    number analyzed (Participants) | 51
    (all) | 262.6 (122.7)
Platelets Level and Neutrophils Level [Mean (Standard Deviation); unit: 10^9 cells per liter] — Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  10^9 cells per liter
    Platelets: number analyzed (Participants) | 60
    Platelets | 260.0 (99.6)
    Neutrophils: number analyzed (Participants) | 58
    Neutrophils | 4.3 (1.6)
Number of Participants Classified According to Heng Prognostic Criteria [Count of Participants; unit: Participants] — Heng prognostic model identified KPS <80 at treatment initiation, period from diagnosis to start of treatment for metastatic disease <1 year, anemia, hypercalcemia, neutrophilia, thrombocytosis as prognostic factors. Participants classified into prognosis group: favorable (0 factor), intermediate (1-2 factors), poor (3 or more factors). KPS measured ability of participants with cancer to perform ordinary tasks. KPS scores range: 0= dead to 100= normal, no complaint. High score= participant better able to carry out daily activities. Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 57
    Favorable | 13
    Intermediate | 40
    Poor | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Remission of Lesions
Description: Time to complete remission of lesions was calculated as the difference between treatment start date and complete response (CR) confirmation date. As per response evaluation criteria in solid tumors (RECIST) version (v) 1.1, CR = disappearance of all known target and all non-target lesions and the absence of new lesions, normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 millimeter (mm). CR was confirmed with 2 consecutive computed tomography (CT) scans performed with at least 4 weeks between them during the follow-up of participants. Confirmation from the oncologist and radiologist was required at each site.
Time Frame: From treatment initiation date to CR confirmation date, up to a maximum of approximately 13 years (from the data collected and observed retrospectively for approximately 10 months)
Population: FAS included all participants who met the inclusion criteria and who did not meet any of the exclusion criteria and received treatment with sunitinib prior to participation in the registry were considered evaluable. This outcome measure was evaluated in participants who achieved CR at respective CT scans.
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 62
Months
  CR at 1st CT Scan | 10.9 [2.4 to 63.2]
  CR at 2nd CT Scan: number analyzed (Participants) | 61
  CR at 2nd CT Scan | 15.7 [5.6 to 67.2]

2. Primary Outcome: Duration of Complete Remission (DOR)
Description: DOR was defined as the time from date on which the CR was identified until tumor progression, the change of treatment due to unacceptable toxicity, death from any cause or until the date of the last follow-up at the close of study. As per RECIST v1.1: CR = disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. Tumor progression = at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of >=5 mm or appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions.
Time Frame: From first documented CR date until progression/death or change of treatment due to unacceptable toxicity or last follow-up date, up to a maximum of approximately 13 years (from the data collected and observed retrospectively for approximately 10 months)
Population: as for outcome 1
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 62
Months
  DOR, 1st CT Scan | 64.1 [6.3 to 145.2]
  DOR, 2nd CT Scan: number analyzed (Participants) | 61
  DOR, 2nd CT Scan | 62.2 [5.3 to 142.5]

3. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was calculated as the time from the date of CR confirmation (2nd CT scan) until the date of progression/death or change of treatment for unacceptable toxicity or censored on the date of the last follow-up. As per RECIST v1.1: CR = disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. Tumor progression = at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of >=5 mm or appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: From CR confirmation date until progression/death or change of treatment due to unacceptable toxicity/last follow-up date, up to maximum of approximately 13 years (data collected, observed retrospectively for approximately 10 months)
Population: FAS included all participants who met the inclusion criteria and who did not meet any of the exclusion criteria and received treatment with sunitinib prior to participation in the registry were considered evaluable.
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 62
Months | NA [NA to NA] — Median and full range could not be estimated because there were insufficient number of participants with event.

4. Other Pre Specified Outcome: Time to Achieve CR in Participants Classified According to Heng I Criteria Prognosis
Description: Time to CR: difference between treatment start date and CR confirmation date. As per RECIST v1.1, CR=disappearance of all known target and all non-target lesions and absence of new lesions, normalization of tumor markers. Pathological lymph nodes must have short axis measures <10mm. CR was confirmed with 2 consecutive CT scans performed with at least 4 weeks between them. Confirmation from oncologist and radiologist was required at each site. Heng prognostic model identified KPS of <80 at treatment initiation, period from diagnosis to start of treatment for metastatic disease <1year, anemia, hypercalcemia, neutrophilia, thrombocytosis as prognostic factors. Participants were classified into 3 prognosis group: favorable(0 factor), intermediate(1-2 factors) and poor(3 or more factors). KPS measured ability of participants with cancer to perform ordinary tasks. KPS scores range: 0 (dead) to 100 (normal, no complaint). High KPS score= participant better able to carry out daily activities.
Time Frame: as for outcome 1
Population: FAS included all participants who met the inclusion criteria and who did not meet any of the exclusion criteria and received treatment with sunitinib prior to participation in the registry were considered evaluable. Here "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies number of participants evaluable for specified rows.
Measure: Median (Full Range); unit: Month
Arm/Group | Sunitinib
Number analyzed (Participants) | 57
Month
  Favorable: number analyzed (Participants) | 13
  Favorable | 9.3 [2.6 to 31.8]
  Intermediate: number analyzed (Participants) | 40
  Intermediate | 11.7 [2.4 to 63.2]
  Poor: number analyzed (Participants) | 4
  Poor | 6.1 [2.8 to 13.5]

5. Other Pre Specified Outcome: Time to Achieve CR in Participants Classified According to Heng I Criteria Prognosis at Least 2 Consecutive CT Scans
Description: Time to CR: difference between treatment start date and CR confirmation date. As per RECIST v1.1, CR=disappearance of all known target and all non-target lesions and absence of new lesions, normalization of tumor markers. Pathological lymph nodes must have short axis measures <10mm. CR was confirmed with 2 consecutive CT scans performed with at least 4 weeks between them. Confirmation from oncologist and radiologist was required at each site. Heng prognostic model identified KPS of <80 at treatment initiation, period from diagnosis to start of treatment for metastatic disease <1year, anemia, hypercalcemia, neutrophilia, thrombocytosis as prognostic factors. Participants were classified into 3 prognosis group: favorable(0 factor), intermediate(1-2 factors) and poor(3 or more factors). KPS measured ability of participants with cancer to perform ordinary tasks. KPS scores range: 0(dead) to 100(normal, no complaint). High KPS score=participant better able to carry out daily activities.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 56
Months
  Favorable: number analyzed (Participants) | 12
  Favorable | 14.8 [7.4 to 37.0]
  Intermediate: number analyzed (Participants) | 40
  Intermediate | 15.5 [5.6 to 67.2]
  Poor: number analyzed (Participants) | 4
  Poor | 10.7 [5.8 to 17.5]

6. Other Pre Specified Outcome: Time to Achieve CR in Participants Classified According to Previous Nephrectomy Status
Description: Time to achieve CR according to previous nephrectomy status were reported in this outcome measure. Time to CR was calculated as the difference between treatment start date and CR confirmation date. As per RECIST v1.1, CR=disappearance of all known target and all non-target lesions and absence of new lesions, normalization of tumor markers. Pathological lymph nodes must have short axis measures <10mm. CR was confirmed with 2 consecutive CT scans performed with at least 4 weeks between them. Confirmation from oncologist and radiologist was required at each site.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 62
Months
  Previous Nephrectomy: Yes: number analyzed (Participants) | 56
  Previous Nephrectomy: Yes | 10.9 [2.4 to 47.2]
  Previous Nephrectomy: No: number analyzed (Participants) | 6
  Previous Nephrectomy: No | 16.6 [6.8 to 63.2]

7. Other Pre Specified Outcome: Time to Achieve CR in Participants Classified According to Histology Type
Description: Time to achieve CR according to type of histology as clear cell, non-clear cell and sarcomatoid were reported in this outcome measure. Time to CR was calculated as the difference between treatment start date and CR confirmation date. As per RECIST v1.1, CR=disappearance of all known target and all non-target lesions and absence of new lesions, normalization of tumor markers. Pathological lymph nodes must have short axis measures <10mm. CR was confirmed with 2 consecutive CT scans performed with at least 4 weeks between them. Confirmation from oncologist and radiologist was required at each site.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 61
Months
  Clear cell: number analyzed (Participants) | 49
  Clear cell | 11.0 [2.4 to 63.2]
  Non-clear cell: number analyzed (Participants) | 5
  Non-clear cell | 8.3 [2.6 to 18.3]
  Sarcomatoid: number analyzed (Participants) | 7
  Sarcomatoid | 9.9 [2.8 to 47.2]

8. Other Pre Specified Outcome: Duration of Response Based on Type of Treatment Received
Description: Duration of response was defined as the time from date on which the CR was identified until the date of the CT scan conforming tumor progression, the change of treatment due to unacceptable toxicity, death from any cause or until the date of the last follow-up at the close of study. As per RECIST v1.1: CR = disappearance of target and non-target lesions and normalization of tumor markers. Pathological lymph nodes must have short axis measures <10 mm. Tumor progression = at least a 20% increase in the sum of diameters of measured lesions taking as references the smallest sum of diameters recorded on study (including baseline) and an absolute increase of >=5 mm or appearance of at least 1 new lesion. Unequivocal progression of existing non-target lesions. Analysis was performed using Kaplan-Meier method.
Time Frame: as for outcome 2
Population: FAS included all participants who met the inclusion criteria and who did not meet any of the exclusion criteria and received treatment with sunitinib prior to participation in the registry were considered evaluable. Here, "number analyzed" signifies number of participants evaluable for specified rows.
Measure: Median (Full Range); unit: Months
Arm/Group | Sunitinib
Number analyzed (Participants) | 62
Months
  Sunitinib Monotherapy: number analyzed (Participants) | 48
  Sunitinib Monotherapy | 69.8 [12.5 to 145.2]
  Sunitinib + subsequent local treatment: number analyzed (Participants) | 14
  Sunitinib + subsequent local treatment | 58.4 [6.3 to 110.1]

9. Other Pre Specified Outcome: Number of Participants With Dose Interruption
Time Frame: From start of drug up to a maximum of approximately 13 years (from the data collected and observed retrospectively for approximately 10 months)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 62
Participants | 47

10. Other Pre Specified Outcome: Number of Participants Who Received Subsequent Local Treatment
Description: Local treatments were the following: traditional surgery, radiotherapy, or stereotactic body radiation therapy (SBRT), to achieve the total macroscopic disappearance of the disease along with CR, according to the opinion of the physician responsible for the participant.
Time Frame: Up to a maximum of approximately 13 years (from the data collected and observed retrospectively for approximately 10 months)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 62
Participants | 14

11. Other Pre Specified Outcome: Number of Participants Who Discontinued Sunitinib Treatment Due to Toxicity
Description: Number of participants who discontinued sunitinib treatment due to toxicity were reported in this outcome measure.
Time Frame: as for outcome 9
Population: FAS included all participants who met the inclusion criteria and who did not meet any of the exclusion criteria and received treatment with sunitinib prior to participation in the registry were considered evaluable. Here "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 34
Participants | 9

12. Other Pre Specified Outcome: Number of Participants With Grade 3 or Higher Toxicity to Sunitinib
Description: Number of participants with Grade 3 or higher toxicity as per common terminology criteria for adverse events (CTCAE) version 4 were reported. Grade 1= mild; Grade 2= moderate; Grade 3= severe; Grade 4= life-threatening or disabling; Grade 5= death.
Time Frame: as for outcome 9
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 51
Participants | 28

ADVERSE EVENTS:
Time Frame: Up to a maximum of approximately 13 years (from the data collected and observed retrospectively for approximately 10 months)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented here are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety set was evaluated. The data collected and observed retrospectively in this study.
Arm/Group | Sunitinib
All-Cause Mortality (participants affected / at risk) | 2/62
Serious Adverse Events (participants affected / at risk) | 9/62
Other Adverse Events (participants affected / at risk) | 51/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=62)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Asthenia (General disorders) | 1
Mucosal inflammation (General disorders) | 2
Bronchitis (Infections and infestations) | 1
Salmonelosis (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=62)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 8
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Cardiotoxicity (Cardiac disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 10
Eyelid oedema (Eye disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 22
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Gastrointestinal toxicity NOS (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 30
Mucosal inflammation (General disorders) | 21
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Conjunctivitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 2
Ejection fraction decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Fluid retention (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyertriglyceridaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 9
Headache (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Albinism (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Hair colour changes (Skin and subcutaneous tissue disorders) | 3
Nail pigmentation (Skin and subcutaneous tissue disorders) | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 25
Rash (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 20
Hypotension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03916458/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/58/NCT03916458/SAP_001.pdf